CLINICAL TRIAL: NCT04778345
Title: Preoperative Abdominal Enhanced CT, 18F-FDG PET/CT and 68Ga-FAPI PET/CT to Detect Peritoneal Carcinomatosis in High-Risk Patients With Gastric Cancer: A Prospective, Single-Center, Comparative Study
Brief Title: Preoperative Abdominal Enhanced CT, 18F-FDG PET/CT and 68Ga-FAPI PET/CT in Peritoneal Carcinomatosis of Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FUGES-021
Record Dates: First submitted 2021-02-22; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Enhanced CT; 18F-FDG PET/CT; 68Ga-FAPI PET/CT; Gastric Cancer; Peritoneal Carcinomatosis
MeSH Terms: conditions — Stomach Neoplasms; Peritoneal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-FDG PET/CT and 68Ga-FAPI PET/CT scan after abdominal enhanced CT (Experimental): After the patient received abdominal enhanced CT, 18F-FDG PET/CT and 68Ga-FAPI PET/CT were further performed. The interval between 18F-FDG PET/CT and 68Ga-FAPI PET/CT was 2 days to 1 week.
  Interventions: Diagnostic Test: 68Ga-FAPI PET/CT scan

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI PET/CT scan — Each subject receives a single intravenous injection of 68Ga-FAPI, and undergo PET/CT imaging after 18F-FDG PET/CT scan during 2 days and 1 week.

SUMMARY:
This study aims to explore the value of 68Ga-FAPI PET/CT in the diagnosis of gastric cancer peritoneal carcinomatosis in high-risk patients compared with conventional abdominal enhanced CT and 18F-FDG PET/CT. The patients with gastric adenocarcinoma (cT4/N+/M0-1) will be studied.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will receive 68Ga-FAPI PET/CT on the 2nd day to 1st week of 18F-FDG PET/CT. On PET/CT, omentum, peritoneum, and mesenteric lesions with increased radioactive uptake are defined as suspicious peritoneal carcinomatosis. The number of these positive lesions, the maximum standardized uptake value (SUVmax), median and range will be recorded. Subsequently, the patients will undergo laparoscopic exploration, and if radical resection is assessed, radical gastrectomy (D2 lymph node dissection) will be performed. If a radical resection is not feasible, for patients with peritoneal carcinomatosis detected, one metastasis will be taken for rapid frozen diagnosis. After the peritoneal carcinomatosis is confirmed, the metastases seen under laparoscopy will be matched with the suspicious peritoneal carcinomatosis on the three preoperative imaging examinations. The intraoperative findings are used as the gold standard to compare the detection efficiency of the three imaging examinations for peritoneal carcinomatosis. Patients with unresected tumors will receive 4 cycles of conversion therapy or neoadjuvant therapy. After the treatment, 18F-FDG PET/CT and 68Ga-FAPI PET/CT will be performed again. If necessary, patients will be subjected to a second laparoscopic exploration, and radical gastrectomy (D2 lymph node dissection) will be performed for appropriate patients. If a radical resection is still not feasible, for patients with peritoneal carcinomatosis detected, biopsy of metastases will be performed if necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 75 years
2. Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
3. The clinical tumor stage before PET/CT scan was evaluated as cT4/N+/M0-1, according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Eighth Edition
4. Performance status of 0 or 1 on Eastern Cooperative Oncology Group scale (ECOG)
5. American Society of Anesthesiology score (ASA) class I, II, or III
6. Written informed consent

Exclusion Criteria:

1. Women during pregnancy or breast-feeding
2. Severe mental disorder
3. History of previous abdominal inflammatory diseases (such as peritonitis, pancreatitis, cholecystitis, inflammatory bowel disease)
4. History of unstable angina or myocardial infarction within past six months
5. History of cerebrovascular accident within past six months
6. History of continuous systematic administration of corticosteroids within one month
7. Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
8. Forced expiratory volume in 1 second (FEV1)<50% of predicted values
9. History of allergy to tracer agents of PET/CT
10. History of allergy to contrast agents of CT

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy for peritoneal carcinomatosis | One month after surgery
  Sensitivity, specificity, accuracy, positive predictive value (PPV) and negative predictive value (NPV) of 68Ga-FAPI PET/CT for peritoneal carcinomatosis in comparison with 18F-FDG PET/CT and abdominal enhanced CT
Maximum standardized uptake value [SUVmax (for PET/CT only)] for peritoneal carcinomatosis | One month after surgery
  SUVmax of 68Ga-FAPI PET/CT for peritoneal carcinomatosis in comparison with 18F-FDG PET/CT

SECONDARY OUTCOMES:
Predictive value for peritoneal carcinomatosis by using radiomic algorithm | One month after surgery
  Prediction value of three kinds of imaging examination for peritoneal carcinomatosis by using radiomic algorithm
Diagnostic efficacy for primary lesions | One month after surgery
  Sensitivity, specificity, accuracy, PPV and NPV of 68Ga-FAPI PET/CT for primary lesions in comparison with 18F-FDG PET/CT and abdominal enhanced CT
SUVmax (for PET/CT only) for primary lesions | One month after surgery
  SUVmax of 68Ga-FAPI PET/CT for primary lesions in comparison with 18F-FDG PET/CT
Diagnostic efficacy for metastatic lymph nodes | One month after surgery
  Sensitivity, specificity, accuracy, PPV and NPV of 68Ga-FAPI PET/CT for metastatic lymph nodes in comparison with 18F-FDG PET/CT and abdominal enhanced CT
SUVmax (for PET/CT only) for metastatic lymph nodes | One month after surgery
  SUVmax of 68Ga-FAPI PET/CT for metastatic lymph nodes in comparison with 18F-FDG PET/CT
Correlation between the expression of fibroblast activation protein (FAP) and 68Ga-FAPI uptake in different pathological types of peritoneal carcinomatosis | One month after surgery
  Analyzing the correlation between the SUVmax of 68Ga-FAPI in peritoneal carcinomatosis with different pathological types and FAP identified by pathological examinations
Correlation between the expression of FAP and 68Ga-FAPI uptake in different pathological types of primary lesions | One month after surgery
  Analyzing the correlation between the SUVmax of 68Ga-FAPI in primary lesions with different pathological types and FAP identified by pathological examinations
Correlation between the expression of FAP and 68Ga-FAPI uptake in different pathological types of metastatic lymph nodes | One month after surgery
  Analyzing the correlation between the SUVmax of 68Ga-FAPI in metastatic lymph nodes with different pathological types and FAP identified by pathological examinations
Predictive value of conversion therapy efficacy | One month after surgery
  Predictive value of three kinds of imaging examination for gastric cancer in conversion therapy response assessment
1-year progression-free survival rate | 12 months
  The relationship between three kinds of imaging examination and the patient's 1-year progression-free survival rate
1-year progression patterns | 12 months
  The relationship between the three types of imaging examinations and the patient's 1-year progression patterns

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Ming Huang, MD, Study Chair — Fujian Medical University Union Hospital
Locations (1):
- Department of Gastric Surgery, Fuzhou, Fujian, China

REFERENCES:
- [Background] Smyth EC, Nilsson M, Grabsch HI, van Grieken NC, Lordick F. Gastric cancer. Lancet. 2020 Aug 29;396(10251):635-648. doi: 10.1016/S0140-6736(20)31288-5. PMID 32861308
- [Background] Roukos DH. Current status and future perspectives in gastric cancer management. Cancer Treat Rev. 2000 Aug;26(4):243-55. doi: 10.1053/ctrv.2000.0164. PMID 10913380
- [Background] Burbidge S, Mahady K, Naik K. The role of CT and staging laparoscopy in the staging of gastric cancer. Clin Radiol. 2013 Mar;68(3):251-5. doi: 10.1016/j.crad.2012.07.015. Epub 2012 Sep 14. PMID 22985749
- [Background] Nakagawa S, Nashimoto A, Yabusaki H. Role of staging laparoscopy with peritoneal lavage cytology in the treatment of locally advanced gastric cancer. Gastric Cancer. 2007;10(1):29-34. doi: 10.1007/s10120-006-0406-3. Epub 2007 Feb 23. PMID 17334715
- [Background] Ajani JA, Bentrem DJ, Besh S, D'Amico TA, Das P, Denlinger C, Fakih MG, Fuchs CS, Gerdes H, Glasgow RE, Hayman JA, Hofstetter WL, Ilson DH, Keswani RN, Kleinberg LR, Korn WM, Lockhart AC, Meredith K, Mulcahy MF, Orringer MB, Posey JA, Sasson AR, Scott WJ, Strong VE, Varghese TK Jr, Warren G, Washington MK, Willett C, Wright CD, McMillian NR, Sundar H; National Comprehensive Cancer Network. Gastric cancer, version 2.2013: featured updates to the NCCN Guidelines. J Natl Compr Canc Netw. 2013 May 1;11(5):531-46. doi: 10.6004/jnccn.2013.0070. PMID 23667204
- [Background] Smyth E, Schoder H, Strong VE, Capanu M, Kelsen DP, Coit DG, Shah MA. A prospective evaluation of the utility of 2-deoxy-2-[(18) F]fluoro-D-glucose positron emission tomography and computed tomography in staging locally advanced gastric cancer. Cancer. 2012 Nov 15;118(22):5481-8. doi: 10.1002/cncr.27550. Epub 2012 May 1. PMID 22549558
- [Background] Garin-Chesa P, Old LJ, Rettig WJ. Cell surface glycoprotein of reactive stromal fibroblasts as a potential antibody target in human epithelial cancers. Proc Natl Acad Sci U S A. 1990 Sep;87(18):7235-9. doi: 10.1073/pnas.87.18.7235. PMID 2402505
- [Background] Hamson EJ, Keane FM, Tholen S, Schilling O, Gorrell MD. Understanding fibroblast activation protein (FAP): substrates, activities, expression and targeting for cancer therapy. Proteomics Clin Appl. 2014 Jun;8(5-6):454-63. doi: 10.1002/prca.201300095. Epub 2014 Mar 24. PMID 24470260
- [Background] Rettig WJ, Su SL, Fortunato SR, Scanlan MJ, Raj BK, Garin-Chesa P, Healey JH, Old LJ. Fibroblast activation protein: purification, epitope mapping and induction by growth factors. Int J Cancer. 1994 Aug 1;58(3):385-92. doi: 10.1002/ijc.2910580314. PMID 7519584
- [Background] Kratochwil C, Flechsig P, Lindner T, Abderrahim L, Altmann A, Mier W, Adeberg S, Rathke H, Rohrich M, Winter H, Plinkert PK, Marme F, Lang M, Kauczor HU, Jager D, Debus J, Haberkorn U, Giesel FL. 68Ga-FAPI PET/CT: Tracer Uptake in 28 Different Kinds of Cancer. J Nucl Med. 2019 Jun;60(6):801-805. doi: 10.2967/jnumed.119.227967. Epub 2019 Apr 6. PMID 30954939
- [Background] Chen H, Pang Y, Wu J, Zhao L, Hao B, Wu J, Wei J, Wu S, Zhao L, Luo Z, Lin X, Xie C, Sun L, Lin Q, Wu H. Comparison of [68Ga]Ga-DOTA-FAPI-04 and [18F] FDG PET/CT for the diagnosis of primary and metastatic lesions in patients with various types of cancer. Eur J Nucl Med Mol Imaging. 2020 Jul;47(8):1820-1832. doi: 10.1007/s00259-020-04769-z. Epub 2020 Mar 28. PMID 32222810
- [Background] Pang Y, Zhao L, Luo Z, Hao B, Wu H, Lin Q, Sun L, Chen H. Comparison of 68Ga-FAPI and 18F-FDG Uptake in Gastric, Duodenal, and Colorectal Cancers. Radiology. 2021 Feb;298(2):393-402. doi: 10.1148/radiol.2020203275. Epub 2020 Dec 1. PMID 33258746
- [Background] Kim JH, Jang YJ, Park SS, Park SH, Kim SJ, Mok YJ, Kim CS. Surgical outcomes and prognostic factors for T4 gastric cancers. Asian J Surg. 2009 Oct;32(4):198-204. doi: 10.1016/S1015-9584(09)60395-X. PMID 19892622
- [Background] Kurita N, Shimada M, Utsunomiya T, Iwata T, Nishioka M, Yoshikawa K, Miyatani T, Higashijima J, Nakao T. Predictive factors of peritoneal metastasis in gastric cancer. Hepatogastroenterology. 2010 Jul-Aug;57(101):980-3. PMID 21033263